CLINICAL TRIAL: NCT05568927
Title: An Observational Cohort Study to Validate SEARCH, a Novel Hierarchical Algorithm to Define Long-term Outcomes After Pulmonary Embolism
Brief Title: Validation of SEARCH, a Novel Hierarchical Algorithm to Define Long-term Outcomes After Pulmonary Embolism
Acronym: ValidSEARCH
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Inari Medical (Industry)
Responsible Party: Principal Investigator, Timothy Morris, Professor of Medicine, University of California, San Diego
Other Study IDs: Inari-RG-2022-01
Record Dates: First submitted 2022-09-28; First posted 2022-10-06 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Embolism; Chronic Thromboembolic Pulmonary Hypertension
Keywords: Clinical validation
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-pulmonary embolism patients: Consecutive patients who, during the study period, underwent the SEARCH algorithm to a diagnostic endpoint at one of the UCAPE network of outpatient pulmonary embolism clinics (UC San Diego, UC Irvine, UC Los Angeles-Harbor, UC Los Angeles, UC Riverside, UC Davis, UC San Francisco or UC San Francisco-Fresno) three months or more after the occurrence of acute pulmonary embolism or any risk type.
  The SEARCH algorithm is the standard of care throughout the UCAPE network, so the experimental portion of this study is limited to the reporting of the (de-identified) results to the evaluation group and the analyses described in Aims 1 and 2. However, there may be patients who are lost to follow up or have other reasons for which the SEARCH algorithm is not followed. Those patients will not be included in the study. The numbers of such patients will be recorded at each center.
  Interventions: Other: SEARCH algorithm

INTERVENTIONS:
Other: SEARCH algorithm — The SEARCH algorithm is a structured, stepwise approach to follow up testing after acute PE that will enable timely diagnosis of post PE sequelae. The test results at each step inform the performance of the subsequent steps. The order of the tests in the algorithm uses the acronym SEARCH: Symptom screen, exercise function, arterial perfusion, resting heart function, confirmatory imaging, and hemodynamics.

SUMMARY:
Potential outcomes after PE occur on a spectrum: complete recovery, exercise intolerance from deconditioning/anxiety, dyspnea from concomitant cardiopulmonary conditions, dyspnea from residual pulmonary vascular occlusion, chronic thromboembolic disease and chronic thromboembolic pulmonary hypertension. Although a battery of advanced diagnostic tests could distinguish each of those conditions, the yield of individual tests among all post- PE patients is low enough that routine testing of all PE patients is not typically performed. Although the various possible post-PE outcomes have enormous implications for patient care, they are rarely distinguished clinically. Perhaps for this reason, chronic conditions after PE are rarely (if ever) used as endpoints in randomized clinical trials of acute PE treatment.

The proposed project will validate a clinical decision tree to distinguish among the various discrete outcomes cost-effectively through a hierarchical series of tests with the acronym SEARCH (for symptom screen, exercise function, arterial perfusion, resting heart function, confirmatory imaging and hemodynamics). Each step of the algorithm sorts a subset of patients into a diagnostic category unequivocally in a cost-effective manner. The categories are mutually exclusive and collectively exhaustive, so that each case falls into one, and only one, category.

Each individual test used in the algorithm has been clinically validated in pulmonary embolism patients, including the cardiopulmonary exercise test (CPET) technique that the investigators developed and validated. However, the decision tree approach to deploying the tests has not yet been validated.

Aim 1 will determine whether the SEARCH algorithm will yield concordant post-PE diagnoses when multiple reviewers independently evaluate multiple cases (reliability).

Aim 2 will determine whether the post-PE diagnoses are stable, according to the SEARCH algorithm, between the first evaluation and the subsequent one six months later (validity).

DETAILED DESCRIPTION:
Study Design Patients with acute pulmonary embolism (PE) receive follow-up care in participating University of California Alliance on Pulmonary Embolism (UCAPE) pulmonary embolism clinics according to the standards of care previously agreed to by the physicians within UCAPE network. At least three months after the onset of acute PE, the patient's physician presents a summary of the case during an on-line meeting without disclosing protected health information or other identifying information. Six designated evaluators independently categorize each patient into a diagnostic endpoint node according to the SEARCH criteria.

SEARCH criteria (positive = at least one criteria met)

Symptoms

* The modified Medical Research Council (mMRC) score on a specific day in the two weeks prior to the interview is one or more points higher than he/she recalls it was on a specific day in the two weeks prior to the PE.
* The patient does not feel fully recovered to the level that existed prior to the PE (e.g. reduced tolerance of athletic abilities), regardless of mMRC scores at the time of the interview and before the PE

Insufficient data: At the first (post-3-month) evaluation, if breathing comfort and exercise tolerance compared to the condition prior to the acute pulmonary embolism could not be ascertained, then the "S" parameter is marked "insufficient data." The patient is excluded from the first primary outcome and the secondary outcome analyses. At the second (6 months subsequent) evaluation, if breathing comfort and exercise tolerance compared to the condition prior to the acute pulmonary embolism could not be ascertained, then the "S" parameter is marked "insufficient data." The patient is be excluded from the second primary outcome and the secondary outcome analyses. If the patient died from pulmonary embolism or pulmonary vascular disease between the first and second evaluations, the patient is to be excluded from the second primary outcome analysis but included in the secondary outcome analyses.If the patient died between the first and second evaluations from a cause other than pulmonary embolism or pulmonary vascular disease, the patient is to be excluded from the second primary outcome and the secondary outcome analyses.

Exercise

* The patient did not reach anaerobic threshold (AT).
* The patient's peak O2 consumption (VO2) was less than (<) 80% of the predicted peak VO2.
* Ventilatory dead space (VD) to tidal volume (VT) ratio (VD/VT) at AT is greater than or equal to (>=) 0.27.
* VD (= VT * VD/VT) in mL at AT is greater than or equal to (>=) 1.35 * the ideal body weight in lbs (IBW).
* In the absence of a VD/VT estimate, the minute ventilation (VE) to CO2 production (VCO2) ratio (VE/VCO2) at AT is greater than (>) 30, which has a sensitivity of 94% and specificity of 48% for a VD/VT at AT greater than 30.
* The ratio of VO2 per heart beat (O2pulse) at AT to the O2pulse at rest (O2pulse_AT/O2pulse_rest) is less than (<) 2.6, which corresponds to stroke volume augmentation at AT of less than 27%.

Insufficient data: At the first evaluation, if S criteria were positive and the patient did not have a subsequent interpretable CPET, then the E parameter is marked "insufficient data." The patient is excluded from the first primary and secondary outcome analyses. At the second evaluation, if S criteria were positive and the patient did not have a subsequent interpretable CPET, then (1) if the S criteria had not worsened since the first time point (mMRC score had not increased), then the results of CPET from the first evaluation point is accepted as true for the second time point; or (2) if the S criteria had worsened (mMRC score increased) and a CPET was not subsequently performed, then the patient is excluded from the second primary outcome and the secondary analysis.

Arterial perfusion

* Planar ventilation: perfusion scanning (planar V:Q) disclosed one or more segmental or larger perfusion defects that do not have matching ventilation defects.
* Planar perfusion scanning (planar Q) disclosed one or more segmental or larger perfusion defects that do not correspond to opacities on chest radiograph or chest CT (performed simultaneously or within 30 days).
* Singe photon emission computer tomography ventilation: perfusion scanning (SPECT V:Q) disclosed one or more segmental or larger perfusion defects that do not have matching ventilation defects.
* SPECT V:Q disclosed one or more segmental or larger perfusion defects that do not correspond to opacities on chest radiograph or chest CT (performed simultaneously or within 30 days).
* The patient did not have an interpretable perfusion scan.

Insufficient data: At the first evaluation, if S and E criteria were positive and the patient did not have a subsequent interpretable perfusion scan, then the A parameter is marked "insufficient data." The patient is excluded from the first primary outcome and the secondary outcome analyses. At the second evaluation, if S and E criteria were positive and the patient did not have a subsequent interpretable perfusion scan, then (1) if the S criteria had not worsened since the first time point (mMRC score had not increased), then the results of the perfusion scan from the first evaluation point is accepted as true for the second time point; or (2) if S criteria had worsened (mMRC score increased) and a perfusion scan was not subsequently performed, then the A parameter is marked "insufficient data." The patient is excluded from the second primary outcome and the secondary analyses.

Resting echocardiography

* Peak tricuspid regurgitation velocity is greater than (>) 2.8 m/s.
* The right ventricle (RV) to left ventricle (LV) ratio (RV/LV) of basal diameters is greater than (>) 1.0.
* There is flattened intraventricular septum or abnormal septal motion.
* Acceleration time of pulmonary ejection is greater than (>) 105 ms or there is midsystolic notching.
* Early diastolic pulmonary regurgitation velocity is greater than (>) 2.2 m/s.
* Pulmonary artery (PA) diameter is greater than (>) 25 mm.
* Tricuspid annular plane systolic excursion (TAPSE) of less than (<) 17 mm.
* Fractional area contraction of RV less than (<) 35% on 4 chamber view.

Insufficient data: At the first evaluation, if S, E and A criteria were positive and the patient did not have a subsequent interpretable echocardiogram, then the R parameter is marked "insufficient data." The patient is excluded from the first primary outcome and the secondary outcome analyses. At the second evaluation, if S, E and A criteria were positive and the patient did not have a subsequent interpretable echocardiogram, then (1) if S criteria had not worsened since the first time point (mMRC score had not increased), then the results of the echocardiogram from the first evaluation point are accepted as true for the second time point; or (2) if S criteria had worsened (mMRC score increased) and an echocardiogram was not subsequently performed, then the R parameter is marked "insufficient data." The patient is excluded from the second primary outcome and the secondary outcome analyses.

Confirmatory imaging

* Smaller than normal caliber arteries contain filling defects
* Eccentric filling defects
* Anastomoses of bronchial arteries
* Right side enlargement
* Contracted lung regions
* Heterogeneous ("mosaic") lung perfusion

Insufficient data: At the first or the second evaluations, absence of interpretable confirmatory imaging (CT or pulmonary angiogram) does not cause the patient to be excluded from the final analysis.

Hemodynamics

* Mean pulmonary artery pressure (mPAP) greater than (>) 20 mmHg with pulmonary arterial wedge pressure less than or equal to (<=) 15 mmHg
* Pulmonary vascular resistance (PVR) greater than or equal to (>=) 3 Wood Units.

Insufficient data: At the first or the second evaluations, absence of right heart catheterization does not cause the patient to be excluded from the final analysis.

X criteria

* During exercise, the mPAP vs cardiac output (CO) slope (mPAP/CO slope) greater than (>) 3 mmHg·L-1·min-1.
* PVR during exercise greater than or equal to (>=) PVR at rest.

Insufficient data: At the first or the second evaluations, absence of right heart catheterization during exercise does not cause the patient to be excluded from the final analysis.

Six months after the first evaluation, the patient's physician presents the case again, along with any updated data, to the UCAPE reader group. Without knowledge of the consensus first evaluation score or the clinically assigned second evaluation score, each member of the UCAPE reader group in the meeting again independently categorizes the patient with a diagnostic endpoint node, using the same on-line scoring tool used for Aim 1. Aim 1 is further described in the Statistics Section under the first and second primary outcomes.

In the instance in which a patient dies after the first evaluation but before the second evaluation could be performed, the patient's physician reviews the case to determine if the death was more likely than not to be related to (1) PE or other pulmonary vascular disease; or (2) an alternative diagnosis.

Aim 2 will determine whether the post-PE diagnoses are stable, according to the SEARCH algorithm, between the first evaluation and the subsequent one (six additional months later). After the scoring procedure described in Aim 1, the mode of the score from the UCAPE readers will be recorded as the consensus score. Aim 2 is further described in the Statistics Section under the secondary outcome.

Quality Assurance

Data Validation

Study facilitators review presentations to ensure lack of protected health information. The presenters validate accuracy of information in the case presentations.

Data checks

A core group performs quality assurance (QA) reviews of test results for completeness, accuracy, uniformity and clarity of (deidentified) data necessary to categorize patients.

Source data verification

Presenters ensure that study data reflects the source data. The presenters will not disclose the patients' identities or any other protected health information to the study staff.

Data dictionary

Pulmonary Embolism - Medical Subject Heading (MeSH) definition Venous Thrombosis - MeSH definition Stroke volume augmentation (SVA): increase in ventricular stroke volume during exercise, compared to stroke volume at rest Physiological dead space proportion (VD/VT): proportion of the ventilatory air in which gas exchange does not occur Chronic thromboembolic disease (CTED): pulmonary hypertension only during exercise due to intravascular pulmonary arterial scars after acute pulmonary embolism Chronic thromboembolic pulmonary hypertension (CTEPH): pulmonary hypertension due to intravascular pulmonary arterial scars after acute pulmonary embolism Symptomatic residual pulmonary vascular occlusion (RPVO): dyspnea or exercise intolerance with objective evidence of segmental or larger mismatched perfusion defects Symptomatic residual pulmonary vascular occlusion with increased VD/VT (RPVO_VD/VT): RPVO with higher-than-normal VD/VT Symptomatic residual pulmonary vascular occlusion with decreased SVA (RPVO_SVA): RPVO with lower-than-normal SVA Symptomatic residual pulmonary vascular occlusion with increased VD and decreased SVA (RPVO_VD+SVA): RPVO with higher-than-normal VD/VT and lower-than-normal SVA Symptomatic residual pulmonary vascular occlusion not otherwise specified (RPVONOS): RPVO with unspecified physiological effect

Standard Operating Procedure Outline

Presenters review all cases in their UCAPE pulmonary embolism follow-up clinics who meet the inclusion criteria. The presenters and a quorum of at least four evaluators independently grade cases.

Missing data

Data that are unavailable, non-reported, uninterpretable, or considered missing because of data inconsistency or out-of-range results will be marked as "missing."

Statistical analysis and sample size estimates

Primary outcome sample size

Fleiss' kappa statistic will measure agreement among the multiple reviewers about the clinical group designation (1-5) for the first evaluation point. The agreement among interpretations will be graded with commonly accepted criteria for kappa values.

Up to six readers review and score cases. Potential outcomes are grouped into five clinically related groups with the following expected probabilities of occurrence:

Symptomatic recovery (59%)

Dyspnea without CPET defects or dyspnea from alternative diagnoses (19%)

Not distinguished among RPVO vs CTED vs CTEPH among RPVO vs CTED vs CTEPH (14%)

RPVO or CTED (13%)

CTEPH (4%).

The expected kappa will be 0.75. With these assumptions, a validation sample set of n = 150 would produce a lower 95% confidence interval (CI) of 0.7 with an alpha of 0.05.

Secondary outcome sample size

For the secondary outcome, we will group the outcomes into six clinically related groups (pi-x), with the sixth group representing death attributed to PE or pulmonary vascular disease:

Symptomatic recovery

Dyspnea without CPET defects or dyspnea from alternative diagnoses or death from alternative diagnoses

Not distinguished among RPVO vs CTED vs CTEPH

RPVO or CTED

CTEPH

Death from PE, CTEPH or other pulmonary vascular disease.

The investigators expect that more than 90% of patients will remain in the same diagnostic group between the first evaluation and the second evaluation. The investigators anticipate that a study size of 150 would disclose 90% agreement and exclude with 95% confidence agreement in fewer than 15% of patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or greater
* objective evidence of acute pulmonary thrombo-embolism at least six months before the evaluation
* anticipated survival for at least three months
* a diagnostic endpoint in the SEARCH algorithm has been reached.

Exclusion Criteria:

● Cases in which the clinical presentations contain insufficient interpretable data to permit evaluation of SEARCH criteria, as described in the Study Design section, will be excluded from the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit consecutive patients who, during the study period, underwent the SEARCH algorithm at one of the UCAPE network of outpatient pulmonary embolism clinics (UC San Diego, UC Irvine, UCLA Harbor, UCLA, UC Riverside, UC Davis, UC San Francisco or UCSF Fresno) three months or more after the occurrence of acute pulmonary embolism or any risk type.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Interobserver agreement among readers regarding the clinical condition during the first evaluation point: at least three months after acute PE. | Each presentation will summarize clinical data leading up to and including an assessment time point at least 3 months after the onset of acute PE
  Based on a structured evaluation of clinical data generated during long term follow-up after PE and presented in a de-identified manner, six observers will independently categorize each patient as one of the following:
  1. complete recovery from dyspnea and exercise intolerance to the state that pre-existed PE or dyspnea after PE but cardiopulmonary exercise test showing normal ventilatory dead space proportions (VD/VT) and normal estimated stroke volume augmentation (SVA) during exercise;
  2. dyspnea after PE likely due to alternative diagnoses;
  3. dyspnea after PE with increased VD/VT or decreased SVA during exercise in the presence of residual pulmonary vascular occlusion (RPVO) but without hemodynamic measurement;
  4. symptomatic RPVO or chronic thromboembolic disease (CTED) documented by hemodynamic measurement;
  5. chronic thromboembolic pulmonary hypertension (CTEPH) documented by hemodynamic measurement.
Interobserver agreement among readers regarding clinical condition at the second evaluation point. | Each presentation will summarize clinical data leading up to and including an assessment time point at least 6 months after the first assessment (described under Aim 1a)
  Based on a structured evaluation of clinical data generated during long term follow-up after PE and presented in a de-identified manner, six observers will independently categorize each patient as one of the following:
  1. complete recovery from dyspnea and exercise intolerance to the state that pre-existed PE or dyspnea after PE but cardiopulmonary exercise test showing normal VD/VT and normal estimated SVA during exercise;
  2. dyspnea after PE likely due to alternative diagnoses;
  3. dyspnea after PE with increased VD/VT or decreased SVA during exercise in the presence of RPVO but without hemodynamic measurement;
  4. symptomatic RPVO or CTED documented by hemodynamic measurement;
  5. CTEPH documented by hemodynamic measurement;
  6. death prior to the evaluation point.

SECONDARY OUTCOMES:
Constancy of diagnosis between first evaluation point and second evaluation point | Stability between the two time points will be determined after the presentation and evaluation of the 12-month time point
  Constancy of diagnosis will be defined as the proportion of patients whose diagnostic category is the same between the first and the second evaluation time points.
  The diagnostic category for the first time point will be the mode of the diagnostic category scores selected by the reviewers among the five options listed for "Outcome 1."
  The diagnostic category for the second time point will be the mode of the diagnostic category scores selected by the reviewers among the six options listed for "Outcome 2."
  Constancy of diagnosis will be calculated as the number of patents with the same diagnoses at the first and second time points divided by the total number of patients who were evaluated at the first and second time points.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Morris, MD, Principal Investigator — University of California, San Diego Healthcare
Locations (8):
- United States (8):
  - University of California, San Francisco-Fresno, Fresno, California
  - University of California, Irvine, Irvine, California
  - University of California, Los Angeles, Los Angeles, California
  - University Hospital, Riverside, Moreno Valley, California
  - University of California, Davis, Sacramento, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of California, Los Angeles - Harbor, Torrance, California

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Background] DeMonaco NA, Dang Q, Kapoor WN, Ragni MV. Pulmonary embolism incidence is increasing with use of spiral computed tomography. Am J Med. 2008 Jul;121(7):611-7. doi: 10.1016/j.amjmed.2008.02.035. PMID 18589057
- [Background] Klok FA, Cohn DM, Middeldorp S, Scharloo M, Buller HR, van Kralingen KW, Kaptein AA, Huisman MV. Quality of life after pulmonary embolism: validation of the PEmb-QoL Questionnaire. J Thromb Haemost. 2010 Mar;8(3):523-32. doi: 10.1111/j.1538-7836.2009.03726.x. Epub 2009 Dec 15. PMID 20025645
- [Background] Klok FA, Tijmensen JE, Haeck ML, van Kralingen KW, Huisman MV. Persistent dyspnea complaints at long-term follow-up after an episode of acute pulmonary embolism: results of a questionnaire. Eur J Intern Med. 2008 Dec;19(8):625-9. doi: 10.1016/j.ejim.2008.02.006. Epub 2008 Apr 22. PMID 19046730
- [Background] Kahn SR, Hirsch AM, Akaberi A, Hernandez P, Anderson DR, Wells PS, Rodger MA, Solymoss S, Kovacs MJ, Rudski L, Shimony A, Dennie C, Rush C, Geerts WH, Aaron SD, Granton JT. Functional and Exercise Limitations After a First Episode of Pulmonary Embolism: Results of the ELOPE Prospective Cohort Study. Chest. 2017 May;151(5):1058-1068. doi: 10.1016/j.chest.2016.11.030. Epub 2016 Dec 6. PMID 27932051
- [Background] Klok FA, van Kralingen KW, van Dijk AP, Heyning FH, Vliegen HW, Kaptein AA, Huisman MV. Quality of life in long-term survivors of acute pulmonary embolism. Chest. 2010 Dec;138(6):1432-40. doi: 10.1378/chest.09-2482. Epub 2010 May 21. PMID 20495104
- [Background] van Es J, den Exter PL, Kaptein AA, Andela CD, Erkens PM, Klok FA, Douma RA, Mos IC, Cohn DM, Kamphuisen PW, Huisman MV, Middeldorp S. Quality of life after pulmonary embolism as assessed with SF-36 and PEmb-QoL. Thromb Res. 2013 Nov;132(5):500-5. doi: 10.1016/j.thromres.2013.06.016. Epub 2013 Oct 3. PMID 24090607
- [Background] Tavoly M, Utne KK, Jelsness-Jorgensen LP, Wik HS, Klok FA, Sandset PM, Ghanima W. Health-related quality of life after pulmonary embolism: a cross-sectional study. BMJ Open. 2016 Nov 3;6(11):e013086. doi: 10.1136/bmjopen-2016-013086. PMID 27810979
- [Background] Kahn SR, Akaberi A, Granton JT, Anderson DR, Wells PS, Rodger MA, Solymoss S, Kovacs MJ, Rudski L, Shimony A, Dennie C, Rush C, Hernandez P, Aaron SD, Hirsch AM. Quality of Life, Dyspnea, and Functional Exercise Capacity Following a First Episode of Pulmonary Embolism: Results of the ELOPE Cohort Study. Am J Med. 2017 Aug;130(8):990.e9-990.e21. doi: 10.1016/j.amjmed.2017.03.033. Epub 2017 Apr 8. PMID 28400247
- [Background] Klok FA, van Kralingen KW, van Dijk AP, Heyning FH, Vliegen HW, Huisman MV. Prospective cardiopulmonary screening program to detect chronic thromboembolic pulmonary hypertension in patients after acute pulmonary embolism. Haematologica. 2010 Jun;95(6):970-5. doi: 10.3324/haematol.2009.018960. Epub 2010 Jan 6. PMID 20053871
- [Background] Fernandes TM, Alotaibi M, Strozza DM, Stringer WW, Porszasz J, Faulkner GG, Castro CF, Tran DA, Morris TA. Dyspnea Postpulmonary Embolism From Physiological Dead Space Proportion and Stroke Volume Defects During Exercise. Chest. 2020 Apr;157(4):936-944. doi: 10.1016/j.chest.2019.10.047. Epub 2019 Nov 22. PMID 31759962
- [Background] Klok FA, van Kralingen KW, van Dijk AP, Heyning FH, Vliegen HW, Huisman MV. Prevalence and potential determinants of exertional dyspnea after acute pulmonary embolism. Respir Med. 2010 Nov;104(11):1744-9. doi: 10.1016/j.rmed.2010.06.006. PMID 20599368
- [Background] Klok FA, Zondag W, van Kralingen KW, van Dijk AP, Tamsma JT, Heyning FH, Vliegen HW, Huisman MV. Patient outcomes after acute pulmonary embolism. A pooled survival analysis of different adverse events. Am J Respir Crit Care Med. 2010 Mar 1;181(5):501-6. doi: 10.1164/rccm.200907-1141OC. Epub 2009 Dec 3. PMID 19965808
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Background] Revicki D, Hays RD, Cella D, Sloan J. Recommended methods for determining responsiveness and minimally important differences for patient-reported outcomes. J Clin Epidemiol. 2008 Feb;61(2):102-9. doi: 10.1016/j.jclinepi.2007.03.012. Epub 2007 Aug 3. PMID 18177782
- [Background] Crisafulli E, Clini EM. Measures of dyspnea in pulmonary rehabilitation. Multidiscip Respir Med. 2010 Jun 30;5(3):202-10. doi: 10.1186/2049-6958-5-3-202. PMID 22958431
- [Background] Kim JW, Clark A, Birring SS, Atkins C, Whyte M, Wilson AM. Psychometric properties of patient reported outcome measures in idiopathic pulmonary fibrosis. Chron Respir Dis. 2021 Jan-Dec;18:14799731211033925. doi: 10.1177/14799731211033925. PMID 34609156
- [Background] Albaghdadi MS, Dudzinski DM, Giordano N, Kabrhel C, Ghoshhajra B, Jaff MR, Weinberg I, Baggish A. Cardiopulmonary Exercise Testing in Patients Following Massive and Submassive Pulmonary Embolism. J Am Heart Assoc. 2018 Mar 3;7(5):e006841. doi: 10.1161/JAHA.117.006841. PMID 29502109
- [Background] McCabe C, Deboeck G, Harvey I, Ross RM, Gopalan D, Screaton N, Pepke-Zaba J. Inefficient exercise gas exchange identifies pulmonary hypertension in chronic thromboembolic obstruction following pulmonary embolism. Thromb Res. 2013;132(6):659-65. doi: 10.1016/j.thromres.2013.09.032. Epub 2013 Sep 27. PMID 24157082
- [Background] Stringer WW, Hansen JE, Wasserman K. Cardiac output estimated noninvasively from oxygen uptake during exercise. J Appl Physiol (1985). 1997 Mar;82(3):908-12. doi: 10.1152/jappl.1997.82.3.908. PMID 9074981
- [Background] Paraskos JA, Adelstein SJ, Smith RE, Rickman FD, Grossman W, Dexter L, Dalen JE. Late prognosis of acute pulmonary embolism. N Engl J Med. 1973 Jul 12;289(2):55-8. doi: 10.1056/NEJM197307122890201. No abstract available. PMID 4710405
- [Background] Prediletto R, Paoletti P, Fornai E, Perissinotto A, Petruzzelli S, Formichi B, Ruschi S, Palla A, Giannella-Neto A, Giuntini C. Natural course of treated pulmonary embolism. Evaluation by perfusion lung scintigraphy, gas exchange, and chest roentgenogram. Chest. 1990 Mar;97(3):554-61. doi: 10.1378/chest.97.3.554. PMID 2106409
- [Background] Donnamaria V, Palla A, Petruzzelli S, Carrozzi L, Pugliesi O, Giuntini C. Early and late follow-up of pulmonary embolism. Respiration. 1993;60(1):15-20. doi: 10.1159/000196167. PMID 8469816
- [Background] Bass H, Banas JS Jr, Dalen JE. Pulmonary function studies. Aid to diagnosis of pulmonary embolism. Arch Intern Med. 1970 Aug;126(2):266-8. doi: 10.1001/archinte.126.2.266. No abstract available. PMID 5433065
- [Background] Sharma GV, Burleson VA, Sasahara AA. Effect of thrombolytic therapy on pulmonary-capillary blood volume in patients with pulmonary embolism. N Engl J Med. 1980 Oct 9;303(15):842-5. doi: 10.1056/NEJM198010093031502. PMID 7412801
- [Background] Helmers RA, Zavala DC. Serial exercise testing in pulmonary embolism. Chest. 1988 Sep;94(3):517-20. doi: 10.1378/chest.94.3.517. PMID 3409730
- [Background] Sanchez O, Helley D, Couchon S, Roux A, Delaval A, Trinquart L, Collignon MA, Fischer AM, Meyer G. Perfusion defects after pulmonary embolism: risk factors and clinical significance. J Thromb Haemost. 2010 Jun;8(6):1248-55. doi: 10.1111/j.1538-7836.2010.03844.x. Epub 2010 Mar 17. PMID 20236393
- [Background] Pesavento R, Filippi L, Palla A, Visona A, Bova C, Marzolo M, Porro F, Villalta S, Ciammaichella M, Bucherini E, Nante G, Battistelli S, Muiesan ML, Beltramello G, Prisco D, Casazza F, Ageno W, Palareti G, Quintavalla R, Monti S, Mumoli N, Zanatta N, Cappelli R, Cattaneo M, Moretti V, Cora F, Bazzan M, Ghirarduzzi A, Frigo AC, Miniati M, Prandoni P; SCOPE Investigators. Impact of residual pulmonary obstruction on the long-term outcome of patients with pulmonary embolism. Eur Respir J. 2017 May 25;49(5):1601980. doi: 10.1183/13993003.01980-2016. Print 2017 May. PMID 28546279
- [Background] Wan T, Rodger M, Zeng W, Robin P, Righini M, Kovacs MJ, Tan M, Carrier M, Kahn SR, Wells PS, Anderson DR, Chagnon I, Solymoss S, Crowther M, White RH, Vickars L, Bazarjani S, Le Gal G. Residual pulmonary embolism as a predictor for recurrence after a first unprovoked episode: Results from the REVERSE cohort study. Thromb Res. 2018 Feb;162:104-109. doi: 10.1016/j.thromres.2017.11.020. Epub 2017 Dec 8. PMID 29224973
- [Background] Pengo V, Lensing AW, Prins MH, Marchiori A, Davidson BL, Tiozzo F, Albanese P, Biasiolo A, Pegoraro C, Iliceto S, Prandoni P; Thromboembolic Pulmonary Hypertension Study Group. Incidence of chronic thromboembolic pulmonary hypertension after pulmonary embolism. N Engl J Med. 2004 May 27;350(22):2257-64. doi: 10.1056/NEJMoa032274. PMID 15163775
- [Background] Leblanc M, Leveillee F, Turcotte E. Prospective evaluation of the negative predictive value of V/Q SPECT using 99mTc-Technegas. Nucl Med Commun. 2007 Aug;28(8):667-72. doi: 10.1097/MNM.0b013e32827a8e99. PMID 17625390
- [Background] Bajc M, Olsson B, Palmer J, Jonson B. Ventilation/Perfusion SPECT for diagnostics of pulmonary embolism in clinical practice. J Intern Med. 2008 Oct;264(4):379-87. doi: 10.1111/j.1365-2796.2008.01980.x. PMID 18823506
- [Background] Lemb M, Pohlabeln H. Pulmonary thromboembolism: a retrospective study on the examination of 991 patients by ventilation/perfusion SPECT using Technegas. Nuklearmedizin. 2001 Dec;40(6):179-86. PMID 11797505
- [Background] Soler X, Hoh CK, Test VJ, Kerr KM, Marsh JJ, Morris TA. Single photon emission computed tomography in chronic thromboembolic pulmonary hypertension. Respirology. 2011 Jan;16(1):131-7. doi: 10.1111/j.1440-1843.2010.01867.x. PMID 20920137
- [Background] Soler X, Kerr KM, Marsh JJ, Renner JW, Hoh CK, Test VJ, Morris TA. Pilot study comparing SPECT perfusion scintigraphy with CT pulmonary angiography in chronic thromboembolic pulmonary hypertension. Respirology. 2012 Jan;17(1):180-4. doi: 10.1111/j.1440-1843.2011.02061.x. PMID 21899658
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Respir J. 2015 Oct;46(4):903-75. doi: 10.1183/13993003.01032-2015. Epub 2015 Aug 29. PMID 26318161
- [Background] Ribeiro A, Lindmarker P, Johnsson H, Juhlin-Dannfelt A, Jorfeldt L. Pulmonary embolism: one-year follow-up with echocardiography doppler and five-year survival analysis. Circulation. 1999 Mar 16;99(10):1325-30. doi: 10.1161/01.cir.99.10.1325. PMID 10077516
- [Background] Ribeiro A, Lindmarker P, Juhlin-Dannfelt A, Johnsson H, Jorfeldt L. Echocardiography Doppler in pulmonary embolism: right ventricular dysfunction as a predictor of mortality rate. Am Heart J. 1997 Sep;134(3):479-87. doi: 10.1016/s0002-8703(97)70085-1. PMID 9327706
- [Background] Remy-Jardin M, Louvegny S, Remy J, Artaud D, Deschildre F, Bauchart JJ, Thery C, Duhamel A. Acute central thromboembolic disease: posttherapeutic follow-up with spiral CT angiography. Radiology. 1997 Apr;203(1):173-80. doi: 10.1148/radiology.203.1.9122389.
- [Background] Cosmi B, Nijkeuter M, Valentino M, Huisman MV, Barozzi L, Palareti G. Residual emboli on lung perfusion scan or multidetector computed tomography after a first episode of acute pulmonary embolism. Intern Emerg Med. 2011 Dec;6(6):521-8. doi: 10.1007/s11739-011-0577-8. Epub 2011 Apr 3. PMID 21461909
- [Background] van Es J, Douma RA, Kamphuisen PW, Gerdes VE, Verhamme P, Wells PS, Bounameaux H, Lensing AW, Buller HR. Clot resolution after 3 weeks of anticoagulant treatment for pulmonary embolism: comparison of computed tomography and perfusion scintigraphy. J Thromb Haemost. 2013 Apr;11(4):679-85. doi: 10.1111/jth.12150. PMID 23347140
- [Background] Hallgren KA. Computing Inter-Rater Reliability for Observational Data: An Overview and Tutorial. Tutor Quant Methods Psychol. 2012;8(1):23-34. doi: 10.20982/tqmp.08.1.p023. PMID 22833776
- [Background] Witten L, Gardner R, Holmberg MJ, Wiberg S, Moskowitz A, Mehta S, Grossestreuer AV, Yankama T, Donnino MW, Berg KM. Reasons for death in patients successfully resuscitated from out-of-hospital and in-hospital cardiac arrest. Resuscitation. 2019 Mar;136:93-99. doi: 10.1016/j.resuscitation.2019.01.031. Epub 2019 Jan 30. PMID 30710595
- [Background] Moskowitz A, Omar Y, Chase M, Lokhandwala S, Patel P, Andersen LW, Cocchi MN, Donnino MW. Reasons for death in patients with sepsis and septic shock. J Crit Care. 2017 Apr;38:284-288. doi: 10.1016/j.jcrc.2016.11.036. Epub 2016 Dec 2. PMID 28013094
- [Background] Sim J, Wright CC. The kappa statistic in reliability studies: use, interpretation, and sample size requirements. Phys Ther. 2005 Mar;85(3):257-68. PMID 15733050
- [Background] Rotondi MA, Donner A. A confidence interval approach to sample size estimation for interobserver agreement studies with multiple raters and outcomes. J Clin Epidemiol. 2012 Jul;65(7):778-84. doi: 10.1016/j.jclinepi.2011.10.019. Epub 2012 May 4. PMID 22560852
- [Derived] Morris TA, Fernandes TM, Chung J, Vintch JRE, McGuire WC, Thapamagar S, Alotaibi M, Aries S, Dakaeva K. Observational cohort study to validate SEARCH, a novel hierarchical algorithm to define long-term outcomes after pulmonary embolism. BMJ Open. 2023 Sep 28;13(9):e074470. doi: 10.1136/bmjopen-2023-074470. PMID 37770267